CLINICAL TRIAL: NCT06372639
Title: Characterization and Modulation of Traumatic Memories in PTSD Patients Using TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Prof., Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAU-PTSD-TMS
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hippocampus Stimulation (Experimental)
  Interventions: Device: Trans-Cranial Magnetic Stimulation
- Sham Stimulation (Sham Comparator)
  Interventions: Device: Trans-Cranial Magnetic Stimulation

INTERVENTIONS:
Device: Trans-Cranial Magnetic Stimulation — Brain stimulation by the TMS device will be given after a deliberate memory re-activation, using repetitive pulses at 1Hz frequency for 15 minutes, the target area will be determined based on an fMRI scan in the resting state of the subject.

SUMMARY:
Characterization and modulation of traumatic memories in PTSD patients using TMS.

DETAILED DESCRIPTION:
Study goals:

1. Characterization of the cortical brain regions that are suitable for effective modulation with TMS, which has the highest connectivity to the sub-cortical regions that are in the strongest connectivity with areas that directly contribute to the formation and preservation of intrusive traumatic memories.
2. Examine the modulation of those cortical brain regions with TMS, while deliberately re-activating an intrusive traumatic memory, on the clinical symptoms of PTSD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20-65 of both sexes, who meet the diagnosis of PTSD according to DSM-5 as tested by a structured clinical interview (Clinician-Administered PTSD Scale - CAPS-5). The clinical interview will be performed by clinical psychologists.
2. CAPS-5 (Clinician-Administered PTSD Scale) score higher than 33.
3. Subjects who experience intrusive symptoms (flashbacks, nightmares, or intrusive memories) at least 4 times a week.
4. Only subjects with a level of Hebrew that allows a full understanding of the consent form to participate in the experiment will be included in the experiment.
5. In addition, the accepted criteria for inclusion for an MRI examination for medical purposes will be applied, according to the established procedures at the MRI Institute at the Sourasky Tel Aviv Medical Center and at the Imaging Center at Tel Aviv University.

Exclusion Criteria:

1. Subjects who meet the diagnosis of Complex PTSD or personality disorder.
2. Subjects who suffer or have suffered in the past from a psychotic disorder, bipolar disorder, or a developmental neuropsychological disorder (autism, mental retardation).
3. Use of psychiatric medications (except for the medications listed in section 4.a) will not be an expense criterion if the medication dosage is stable in the last three months and does not change during the study.

   In addition, exclusion criteria 4-13 will apply according to the exclusion rules in TMS laboratories in England and the USA:
4. Use of the following drugs:

   a. The list of drugs that constitute a criterion for exclusion in the study: imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, (MDMA, ecstasy), phencyclidine (PCP, angel's dust), ketamine, gamma- hydroxybutyrate (GHB), alcohol, theophylline
5. Subjects suffering from epilepsy or taking anti-epileptic drugs.
6. Victims with traumatic head injuries or who have undergone head surgery.
7. Having a metallic body (except fillings/amalgam bites/orthodontic fixations approved for MRI), electrodes or a pacemaker in their body.
8. Subjects suffering from migraines
9. Pregnant women
10. Subjects with hearing problems
11. Subjects who use drugs
12. Subjects who drank alcohol 24 hours before the experiment
13. Subjects who have previously experienced repeated episodes of fainting with loss of consciousness and/or an event of fainting with loss of consciousness in the past year. (reaction and vegalit)
14. In addition, the accepted exclusion criteria for an MRI examination for medical purposes will apply, according to the established procedures at the MRI Institute at the Sourasky Tel Aviv Medical Center and at the Imaging Center at Tel Aviv University.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
CAPS-5 score | Baseline, second measure after up to 12 weeks and last measure after up to 24 weeks.
  The CAPS-5 is a 30-item structured interview that can be used to make current (past month or week) diagnosis of PTSD & make lifetime diagnosis of PTSD.
Neurological measures of functional connectivity | Baseline, after up to 12 weeks
  Functional connectivity, indicating the level of synchronous activity of certain brain regions during rest (temporal correlation is usually expressed as a Pearson's r); Also to be derived from the MRI scans, and compared between the two groups over time.
Intrusive memories | Daily for up to 12 weeks
  The amount, frequency and emotional effect of intrusive traumatic memories, measured by a daily self-report of the subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel